CLINICAL TRIAL: NCT04600544
Title: Disease-oriented Russian Disc Degeneration Study (RuDDS) Biobank Facilitating Functional Omics Studies of Lumbar Disc Degeneration
Brief Title: Russian Disc Degeneration Study
Acronym: RuDDS
Status: Completed | Type: Observational
Sponsor: Novosibirsk State University (Other)
Collaborators: Institute of Cytology and Genetics (Unknown); Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan (Other Government); N.N. Priorov National Medical Research Center of Traumatology and Orthopedics (Other)
Responsible Party: Sponsor
Other Study IDs: NS02-04
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Intervertebral Disc Degeneration; Genetic Predisposition to Disease
Keywords: biobank; functional genomics; transcriptomics; glycomics
MeSH Terms: conditions — Intervertebral Disc Degeneration; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Whole blood samples, plasma. Intervertebral lumbar disc samples only for patients subjected for surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional — Translational, observational study

SUMMARY:
The main aim of this study is to establish disease-oriented biobank to facilitate research in biology of the lumbar disc degeneration. Diverse biological samples (whole blood, plasma, disc tissue) along with MRI imaging, clinical, socio-demographic and various omics data (e.g. genomic and transcriptomic) will be available for researchers and clinicians for a variety of further multi-omics studies. It will lay the groundwork for the development of early diagnostics of DDD and its personalized treatment.

The study is planned to enroll up to 1,100 patients with different grades of lumbar disc degeneration. It is planned to recruit patients within 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18;
2. Presence of lumbar MRI scans;
3. Signed informed consent for voluntary participation is provided.

Exclusion Criteria:

1. Any contraindication or inability to undergo baseline procedures;
2. Prior surgeries at any level of the lumbar spine;
3. Other non-degenerative spinal conditions that may have an impact on subject safety, wellbeing or the intent and conduction of the study;
4. History or presence of HIV, hepatitis B, hepatitis C.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants aged over 18 with available MRI scans of lumbar spine, who will also sign an informed consent and meet all the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1070 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Genotyping | Through 3 years
  DNA will be extracted from the whole blood samples according to the standard protocol

SECONDARY OUTCOMES:
Phenotype of patients with lumbar disc degeneration | Through 3 years
  General information about a patient, his medical history and MRI scans of lumbar spine
Total plasma proteins N-glycosylation profiling | Through 3 years
  The plasma glycans profiling will be performed according to standard protocol
Total RNA profiling | Through 3 years
  The intraoperative material will be homogenized and total RNA will be extracted and converted to cDNA using Kit for the isolation of total RNA and microRNA from cells and tissues and M-MuLV-RH First Strand cDNA Synthesis Kit respectively. The amount of extracted RNA and its quality will be estimated using Bioanalyzer 2100.

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Priorov National Medical Research Center of Traumatology and Orthopedics, Moscow
  - Institute of Cytology and Genetics, Novosibirsk
  - Novosibirsk Research Institute of Traumatology and Orthopaedics n.a.Ya.L.Tsivyan, Novosibirsk

IPD SHARING:
Plan to Share IPD: Yes
To access the database, omcis data and other relevant information, projects should be submitted to the steering committee (contact the Central Contact Person) of the RuDDS.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: During the study conducting and 5 years after
Access Criteria: Contact the Central Contact Person onleonova@gmail.com

REFERENCES:
- [Derived] Leonova O, Elgaeva E, Berdnikova A, Tsepilov Y, Krutko A. Lumbar MRI and Back Pain After Failed Conservative Treatment: The RuDDS Study. Global Spine J. 2025 Sep 3;16(2):21925682251373046. doi: 10.1177/21925682251373046. Online ahead of print. PMID 40901806
- [Derived] Leonova ON, Elgaeva EE, Golubeva TS, Peleganchuk AV, Krutko AV, Aulchenko YS, Tsepilov YA. A protocol for recruiting and analyzing the disease-oriented Russian disc degeneration study (RuDDS) biobank for functional omics studies of lumbar disc degeneration. PLoS One. 2022 May 13;17(5):e0267384. doi: 10.1371/journal.pone.0267384. eCollection 2022. PMID 35560143